CLINICAL TRIAL: NCT05483140
Title: Assessing The Effectiveness of A Digitally Enabled Low Energy Diet on Type 2 Diabetes Management
Brief Title: Digitally-Enabled Weight Management Program on T2DM
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Collaborators: Changing Health (Unknown); National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: HA55
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Weight Change, Body; Type 2 Diabetes
MeSH Terms: conditions — Body Weight Changes; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low Energy Diet Group: A low energy diet comprising of three options and lifestyle modifications as part of a digitally enabled weight loss program.
  Interventions: Other: Option 1; Other: Option 2; Other: Option 3

INTERVENTIONS:
Other: Option 1 — Partial meal replacement to achieve 900-1000 kcal/day (4 meal replacement products per day combined with 150-200 kcal from vegetable meals (recipes provided))
Other: Option 2 — Partial meal replacement to achieve 900-1000 kcal/day (2 meal replacement products per day combined with one balanced meal (recipes provided))
Other: Option 3 — A real food low energy diet to achieve 800-1000 kcal/day (recipes provided)

SUMMARY:
The study (known as clinical audit in UK) will observe and report on a digitally-enabled structured weight management program including use of a meal replacement on clinical and economic outcomes for community-dwelling adults living with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Have a clinical diagnosis of T2DM within the last 6 years
2. Aged 20 - 70 years
3. Have a BMI ≥ 27 kg/m2
4. HbA1c ≥ 48 mmol/mol (≥ 42mmol/mol if prescribed glucose-lowering agents)
5. Have access to the internet and a computer, smartphone or tablet
6. Ability to read and understand English
7. Willing to provide individual consent

Exclusion Criteria:

1. Current insulin use
2. More than two anti-hyperglycemic agents prescribed
3. Recent routine HbA1c ≥ 90 mmol/mol
4. Diagnosed with moderate or severe frailty
5. Diagnosed eating disorder or purging
6. Unable or unwilling to tolerate soy/milk-based meal replacements
7. Myocardial infarction within last 6 months
8. Recent eGFR <30 ml/min/1.73 m2
9. Prescribed SGLT2 inhibitor for diabetic kidney disease (DKD) or left ventricular hypertrophy (LVH)
10. Severe heart failure defined as equivalent to the New York Heart Association grade 3 (NYHA)
11. Current treatment with anti-obesity drugs
12. Learning difficulties that would prevent engagement with the program
13. Having required hospitalization for depression or being prescribed antipsychotic drugs
14. Known cancer
15. Active substance misuse
16. Contraindications to exercise
17. Contraindications to lose weight
18. Mental or physical incapacity that makes self-management inappropriate
19. Pregnant, planning a pregnancy or lactating
20. Currently undergoing palliative care
21. Previous bariatric surgery or on waiting list for bariatric surgery (unless willing to come off waiting list)
22. Unable to commit to long term lifestyle change
23. Known proliferative retinopathy that has not been treated

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community-dwelling adults - In partnership with North East and North Cumbria NHS Integrated Care System (ICS) we will engage with the four integrated care providers (ICP) and their Primary Care Networks (PCNs) across this system to identify and receive eligible referrals for participation in this program
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Program Feasibility | Baseline to 12 Months
  Participant and HCP completed program questionnaire scored from 0 to 10 where higher score is more favorable
Program Effectiveness | Baseline to 12 Months
  Mean Weight Change

SECONDARY OUTCOMES:
Glycemic Control | Baseline to 12 Months
  Mean HbA1c change
Diabetes Distress | Baseline to 12 Months
  Participant completed PAID5 (Problem Areas In Diabetes) diabetes-related emotional distress scale from 0 to 100 where higher rating is less favorable
Medication Usage use | Baseline to 12 Months
  Medications prescribed from baseline throughout study phases

OTHER OUTCOMES:
Healthcare Resource Utilization (HRU), including unplanned (non-study-related) (re)hospitalizations, emergency department (ED) visits, and outpatient clinic visits, depending on data | Baseline to 12 Months
  Number of unplanned inpatient hospitalizations, outpatient clinic visits, emergency department visits
HRU Cost-Savings service, depending on data availability. | Baseline to 12 Months
  Change in cost of overall healthcare resource utilization
Quality of Life (QOL) SF-12 | Baseline to 12 Months
  Patient Reported (QOL) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Maria Camprubi, PhD, Study Chair — Abbott Nutrition
Locations (4):
- United Kingdom (4):
  - Nhs Tees Valley Ccg, Middlesbrough
  - Nhs Northumberland Ccg, Morpeth
  - Nhs Newcastle Gateshead Ccg, Newcastle upon Tyne
  - Nhs North Tyneside Ccg, North Shields

IPD SHARING:
Plan to Share IPD: No